CLINICAL TRIAL: NCT00003484
Title: Phase I Study of Anti-Tenascin Monoclonal Antibody I-Labeled 81C6 Via Surgically Created Cystic Resection Cavity in the Treatment of Patients With Primary Brain Tumors After External Beam Radiotherapy
Brief Title: Radiolabeled Monoclonal Antibody Therapy After Radiation Therapy in Treating Patients With Primary Brain Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Darell D. Bigner, MD, PhD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Darell D. Bigner, MD, PhD, Director, The Preston Robert Tisch Brain Tumor Center at Duke, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00008915; DUMC-1533-02-8R5ER (Other: Duke University IRB); DUMC-1533-01-8R4 (Other: Duke University IRB); DUMC-1373-97-9 (Other: Duke University IRB); DUMC-1408-98-9R1 (Other: Duke University IRB); DUMC-1533-00-8R3 (Other: Duke University IRB); DUMC-1570-99-9R2 (Other: Duke University IRB); DUMC-97107 (Other: Duke University Cancer Protocol Committee); 5P0NS20023 (Other Grant/Funding Number: National Cancer Institute); NCI-G98-1472 (Other Grant/Funding Number: National Cancer Institute); CDR0000066522 (Other: National Cancer Institute Record Identifier)
Record Dates: First submitted 1999-11-01; First posted 2003-04-30 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Brain and Central Nervous System Tumors; Neuroblastoma
Keywords: localized resectable neuroblastoma; recurrent adult brain tumor; adult craniopharyngioma; adult medulloblastoma; adult meningioma; adult glioblastoma; adult oligodendroglioma; adult anaplastic astrocytoma; adult mixed glioma; adult pineal parenchymal tumor; adult central nervous system germ cell tumor; adult grade III meningioma; adult pilocytic astrocytoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Neuroblastoma; Brain Neoplasms; Craniopharyngioma; Medulloblastoma; Meningioma; Glioblastoma; Oligodendroglioma; Astrocytoma; Glioma; Pinealoma; Gliosarcoma | interventions — Carmustine; Irinotecan; Surgical Procedures, Operative

INTERVENTIONS:
Drug: carmustine
Drug: irinotecan hydrochloride
Procedure: surgical procedure
Radiation: iodine I 131 monoclonal antibody 81C6

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and deliver tumor-killing substances, such as radioactive iodine, to them without harming normal cells.

PURPOSE: Phase I trial to study the effectiveness of radiolabeled monoclonal antibody after radiation therapy in treating patients with newly diagnosed primary brain tumors that can be surgically resected.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity of iodine I 131 monoclonal antibody 81C6 delivered via the intracranial resection cavity in patients with newly diagnosed primary malignant brain tumors after surgery and radiotherapy.
* Determine objective therapeutic responses of these patients to this treatment.

OUTLINE: This is a dose escalation study of iodine I 131 antitenascin monoclonal antibody 81C6 (I 131 MAb 81C6).

Within 2-4 weeks after completion of external beam radiotherapy, patients undergo surgical resection of the tumor or brain metastasis, at which time an indwelling intracranial resection cavity catheter is placed. A single dose of I 131 MAb 81C6 is delivered via the intralesional catheter.

Cohorts of 3-6 patients receive escalating doses of I 131 MAb 81C6 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicities.

After the MTD has been established, patients in the phase II portion of the study receive therapy as in phase I.

Beginning 4 weeks after the monoclonal antibody treatment, patients begin chemotherapy. Patients receive carmustine IV over 1 hour on day 1 and irinotecan IV over 90 minutes once weekly for 4 weeks. Treatment is repeated every 6 weeks for at least 4 courses in the absence of disease progression.

Patients are followed initially at 4 weeks, then every 6 weeks for 1 year.

PROJECTED ACCRUAL: A total of 41 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed newly diagnosed supratentorial primary malignant brain tumor
* No infratentorial tumors, infiltrating tumors, tumors with subependymal spread, or multifocal tumors
* Candidate for surgical resection
* Prior external beam radiotherapy to site of measurable disease or resection site in the nervous system required
* Presence of tenascin in the tumor demonstrated by immunohistology with either a polyclonal rabbit antitenascin antibody or monoclonal antibody 81C6

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 50-100%

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count greater than 1000/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin less than 1.5 mg/dL
* Alkaline phosphatase less than 1.5 times normal
* Lactic dehydrogenase less than 1.5 times normal
* SGOT less than 1.5 times normal

Renal:

* Creatinine less than 1.2 mg/dL

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No iodine allergies

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Concurrent corticosteroids allowed, but must be on stable dose for at least 10 days

Radiotherapy:

* See Disease Characteristics

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 1997-09; Primary Completion 2003-11 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darell D. Bigner, MD, PhD, Study Chair — Duke University
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States